CLINICAL TRIAL: NCT06233123
Title: Efficacy of a Phone Application on Treatment Adherence in Asthmatic Patients in Upper Egypt
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Entsar Hsanen, doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: asthma adherence phone
Record Dates: First submitted 2024-01-12; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Bronchial Asthma; Adherence, Medication
MeSH Terms: conditions — Asthma; Medication Adherence | interventions — Artificial Intelligence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Application (Experimental): intervention group that will download the Medisafe android application (https://www.medisafe.com). This mobile application uses simple English language and figures to remind the patient about the dose
  Interventions: Behavioral: the Medisafe android application (https://www.medisafe.com).
- control (No Intervention): control group with Standard Care and Medication Monitoring

INTERVENTIONS:
Behavioral: the Medisafe android application (https://www.medisafe.com). — software for Android mobile phones that can remind the patient of his treatment on time
  Other Names: Artificial intelligence; mobile application; phone application
  Arms: Application

SUMMARY:
asthma adherence is mandatory for disease control

DETAILED DESCRIPTION:
Asthma is a chronic and common disease of the airways that affects more than 339 million people globally [1]. According to WHO estimates, there were 417,918 deaths due to asthma at the global level and 24.8 million disability-adjusted life years (DALYs) attributable to Asthma [2, 3]. There is much evidence that self-care by patients with asthma has beneficial outcomes, including reduced hospital stays, reduced symptoms, and general compliance with treatments [4-6]. One of the approaches for promoting self-care skills in patients with asthma is to provide self-care services (i.e., providing basic information about the nature of asthma, avoiding exposure to allergens and triggers, treating with drugs, providing alerts and reminders to patients, and how to use the therapeutic tools [7]) through information technology tools (e.g. the Internet, mobile phones, and computer software). Given the increasing worldwide use of smartphones, mobile health (mHealth) technologies can work as promising tools to improve self-care in patients with asthma by providing support services such as communication information, providing learning materials, and sending reminders for behavior change [8, 9]. mHealth, as a component of electronic health, is related to the use of mobile phones and other wireless technologies to improve the provision of health-related services. Moreover, ease of use, portability, and ubiquity in all regions are the potential benefits of mHealth tools for the prevention, diagnosis, treatment, and care of diseases also increasing access to health services and reducing the costs incurred [10]. This study aims to evaluate the role of a mobile application in reminding the patient to take his treatment and its reflection on asthma control and quality of life.

ELIGIBILITY:
Inclusion Criteria:

Doctor-diagnosed asthma. On at least Global Initiative for Asthma (GINA) step 3 which means they will be on regular inhaled steroids.

No change in regular asthma treatment in the last 1 month Sufficient English-language ability to understand the text in mobile phone-delivered interventions The education level required will be at least a high school diploma.

Exclusion Criteria:

GINA step 5 asthma (complex issues, too unstable). Recent changes to asthma treatment within the last month Another chronic health condition (eg diabetes, congenital heart disease, cystic fibrosis) Patients without mobile device skills

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Asthma control after 3 months | 3 months
  asthma control test after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Entsar H Mohamed, Lecturer, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Vos T, Abajobir AA, Abate KH, et al. Global, regional, and national incidence, prevalence, and years lived with disability for 328 diseases and injuries for 195 countries, 1990-2016: a systematic analysis for the Global Burden of Disease Study 2016. The Lancet. 2017;390(10100):1211-59. 2.World Health Organisation. Global health estimates 2016: deaths by cause, age, sex, by country and by region, 2000-2016. Geneva: World Health Organization; 2018a. 3.World Health Organisation. Global health estimates 2016: disease burden by cause, age, sex, by country and by region, 2000-2016. Geneva: World Health Organization; 2018b. 4.Levy M, Andrews R, Buckingham R, et al. Why asthma still kills: the National Review of Asthma Deaths (NRAD). London: Royal College of Physcians; 2014. 5.James DR, Lyttle MD. British guideline on the management of asthma: SIGN Clinical Guideline 141, 2014. Arch Dis Child Educ Pract. 2016;101(6):319-22.
- Available data/document: Individual Participant Data Set — https://pubmed.ncbi.nlm.nih.gov/32021311/